CLINICAL TRIAL: NCT04314700
Title: Intraoperative Use of the OTIS™ (OCT Imaging System) to Guide Additional Margin Cavity Shaves in Breast Conserving Surgery (BCS)
Brief Title: Intraoperative Use of an Optical Coherence Tomography (OCT) Imaging System to Guide Additional Margin Cavity Shaves in Breast Conserving Surgery (BCS)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the site
Sponsor: Perimeter Medical Imaging (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: PER-19-02
Record Dates: First submitted 2020-03-03; First posted 2020-03-19 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- OCT imaging and review of excised breast lumpectomy tissue (Other)
  Interventions: Device: OCT- based investigational imaging device

INTERVENTIONS:
Device: OCT- based investigational imaging device — Excised breast lumpectomy tissue will be imaged and images reviewed on an investigational Wide-Field OCT (WF-OCT) device.

SUMMARY:
Female patients undergoing a breast conserving procedure will be consented for the excised breast tissue to be imaged on an investigational OCT-based device. Additional tissue may be excised to obtain clear/negative margins based on routine standard of care tissue assessment techniques and intraoperative OCT image review.

DETAILED DESCRIPTION:
Note: A retrospective review of the stated purpose and objectives of the PER-19-02 protocol has determined that this study better fits the definition of a medical device feasibility study, with regard to FDA guidance "Investigational Device Exemptions (IDEs) for Early Feasibility Medical Device Clinical Studies, Including Certain First in Human (FIH) Studies," issued October 2013. The primary objectives of the PER-19-02 study (NCT04314700) emphasize user factors, rather than health outcomes, as the focus is on collecting information related to usability and timing, with no change to the standard of care (pathology analysis and additional surgery when needed). PER-19-02 was not used as a pivotal study to support the substantial equivalence or safety and effectiveness evidence submitted as part of an FDA pre-market submission. The IDE-approved pivotal study for evaluating the effect of Perimeter's OCT technology on health-related outcomes in breast surgery is the randomized control trial registered on ClinicalTrials.gov under protocol PER-19-04 (NCT05113927). Perimeter has determined this trial does not meet the definition of an Applicable Clinical Trial per the "Checklist for Evaluating Whether a Clinical Trial or Study is an Applicable Clinical Trial (ACT) Under 42 CFR 11.22(b) for Clinical Trials Initiated on or After January 18, 2017."

ELIGIBILITY:
Inclusion Criteria:

* Female age 18 or older
* Patients undergoing elective breast conservation surgery for the treatment of Stage 0-III invasive ductal or lobular breast carcinoma and/or ductal carcinoma in situ
* May include subjects treated with neo-adjuvant endocrine therapy
* May include subjects treated with neo-adjuvant chemotherapy with confirmed complete clinical response
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Male
* Stage IV breast cancer
* Participation in another study that prolongs time to pathologic processing (greater than 1 hour)
* Neo-adjuvant treated patients with any chemotherapeutic who have not achieved a complete clinical response
* A surgeon makes an intraoperative decision to conduct a frozen section analysis (Any subject-specific data collected from an enrolled subject until the surgeon's intraoperative decision will not be used in the data analysis of this study. These subjects will be replaced in the study and the surgeon's intraoperative decision to conduct a frozen section analysis will be recorded).
* Use of cryosurgery
* Currently lactating
* Current pregnancy
* Previous ipsilateral breast surgery for benign or malignant disease in the same quadrant as currently planned surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
Number of times the surgeon recorded a decision to excise additional tissue based on intra-operative Wide Field Optical Coherence Tomography (WF-OCT) image review in addition to Standard of Care tissue assessment. | Within 1 hour of tissue excision
  Surgeon's assessment of margin status post Wide Field OCT (WF-OCT) image review and any action taken, will be recorded.
Average time to excise additional tissue during Breast Conserving Surgery (BCS) | Within 1 hour of primary tumor excision
  Time taken to excise additional tissue based on WF-OCT image review, will be recorded.
Calculate percentage of patients that require a second surgery | Within about 3 months of first surgery
  Record percentage of patients with positive margins per pathology, that require a second surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Beth DuPree, MD, Principal Investigator — Northern Arizona Healthcare
Locations (1):
- Northern Arizona Healthcare, Cottonwood, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified Individual Participant Data (IPD) may be shared with other researchers and the sponsor for research/product development purposes.
Supporting Information: Study Protocol, CSR
Time Frame: During the study and post study completion
Access Criteria: Research and development/product development purposes.